CLINICAL TRIAL: NCT00574665
Title: SCCOR in Hemostatic and Thrombotic Diseases Project 5 - Metabolic Causes of Thrombosis in Type 2 Diabetes
Brief Title: Metabolic Causes of Thrombosis in Type 2 Diabetes - Question 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steve Davis, Department Chair, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#060227-SCCOR-Q1; RFAHL04016
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Endothelial Function; Fibrinolytic Balance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Hyperinsulinemic Hyperglycemic Clamp

INTERVENTIONS:
Other: Hyperinsulinemic Hyperglycemic Clamp — Glucose Clamp

SUMMARY:
The purpose of this study is to learn more about why patients with diabetes have increased heart attacks, strokes and other illnesses due to blood clots causing blockage of a blood vessel. The proposed protocol will study the separate and combined effects of hyperglycemia and hyperinsulinemia on endothelial function and fibrinolytic balance in Type 2 DM. Our hypothesis is that hyperglycemia, rather than hyperinsulinemia, is responsible for the dysregulation of fibrinolytic balance in diabetics.

DETAILED DESCRIPTION:
This study will test the hypothesis that hyperglycemia will impair, while hyperinsulinemia will improve endothelial function and vascular fibrinolytic balance in type 2 DM. As discussed above, their roles in the increased prevalence of thrombotic events occurring in diabetics have not been defined. More recent data supports insulin as profibrinolytic and hyperglycemia to cause endothelial dysfunction. Conclusive studies are lacking in diabetic subjects. Furthermore, preliminary data from this lab indicates that in non-diabetic controls, hyperglycemia results in a prothrombotic state by increasing plasma PAI-1 and reducing tPA levels. The proposed protocol will study the separate and combined effects of hyperglycemia and hyperinsulinemia on endothelial function and fibrinolytic balance in Type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* 16 ( 8 female/ 8 male) Type 2 diabetic patients age 18-60 yrs
* 16 ( 8 female/ 8 male) Non-diabetic controls age and weight matched
* Body mass index 25-52 kgm2
* Female volunteers of childbearing potential: negative HCG pregnancy test
* Volunteers over 40 years old: normal baseline ECG
* For those with type 2 diabetes: HBA1C 6.5-10%

Exclusion Criteria:

* Prior history of poor health: any current or prior disease condition that alters carbohydrate metabolism and prior cardiac events and/or evidence for cardiac disease
* Uncontrolled hypertension
* History of cerebrovascular incidents
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with a recent medical illness
* Subjects with known liver or kidney disease
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases
* Tobacco Use

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function and fibrinolytic balance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States